CLINICAL TRIAL: NCT04253847
Title: Radical Antegrade Modular Pancreatosplenectomy Versus Standard Retrograde Pancreatosplenectomy on the Survival and Prognosis for Resectable Body and Tail Pancreatic Ductal Adenocarcinoma
Brief Title: RAMPS VS SRPS for Pancreatic Body and Tail Adenocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yuanchi Weng, Attending Physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBP-RCT-005
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Radical Antegrade Modular Pancreatosplenectomy
Keywords: Radical antegrade modular pancreatosplenectomy; Standard retrograde pancreatosplenectomy; Pancreatic Body and Tail Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will not know which group they are assigned to, but the surgeons know which group they were randomly assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAMPS group (Experimental): Radical antegrade modular pancreatosplenectomy (RAMPS) includes the following aspects. Firstly, the surgical approach is "antegrade", which means from the right to the left, the pancreatic neck will be transected at first and the spleen will be seperated at last. Secondly, lymph nodes dissection includes not only the regional lymph nodes(No.10,11,18 lymph nodes), but also N1 station lymph nodes (N1: 6, 8a, 8p, 12a2/b2/p2, 13a/b, 14b/c/d, 14v, 17a/b), No.7, 9 lymph nodes, the lymph nodes anterior and left of superior mesenteric artery, as well as the peripheral nerve of celiac trunk. Thirdly, the transection platform is in the pancreatic neck, which is mandatory. At last, left prerenal fascia will be resected. When the tumor abuts or infiltrates the left adrenal gland, left adrenalectomy will be performed, which is also called "posterior approach RAMPS". While in normal cases, left adrenal gland will be preserved.
  Interventions: Procedure: Radical antegrade modular pancreatosplenectomy
- SRPS group (Active Comparator): Standard retrograde pancreatosplenectomy(SRPS) includes several key points. Firstly, the surgical approach is "retrograde", which means from the left to the right, spleen will be seperated at first and the pancreas will be transected later on. Secondly, only the regional lymph nodes will be dissected, which include No.10, No.11, No.18 lymph nodes, and No.9 lymph nodes should be dissected only when the lesion is in pancreatic neck. Thirdly, the transection platform is in the left side of the lesion, but transection at pancreatic neck is not mandatory. At last, the surgical plane is anterior to the left renal fascia, prerenal fascia will be preserved.
  Interventions: Procedure: Standard retrograde pancreatosplenectomy

INTERVENTIONS:
Procedure: Radical antegrade modular pancreatosplenectomy — Radical antegrade modular pancreatosplenectomy (RAMPS) includes the following aspects. Firstly, the surgical approach is "antegrade", which means from the right to the left, the pancreatic neck will be transected at first and the spleen will be seperated at last. Secondly, lymph nodes dissection includes not only the regional lymph nodes(No.10,11,18 lymph nodes), but also N1 station lymph nodes (N1: 6, 8a, 8p, 12a2/b2/p2, 13a/b, 14b/c/d, 14v, 17a/b), No.7, 9 lymph nodes, the lymph nodes anterior and left of superior mesenteric artery, as well as the peripheral nerve of celiac trunk. Thirdly, the transection platform is in the pancreatic neck, which is mandatory. At last, left prerenal fascia will be resected. When the tumor abuts or infiltrates the left adrenal gland, left adrenalectomy will be performed, which is also called "posterior approach RAMPS". While in normal cases, left adrenal gland will be preserved.
  Arms: RAMPS group
Procedure: Standard retrograde pancreatosplenectomy — Standard retrograde pancreatosplenectomy(SRPS) includes several aspects. Firstly, the surgical approach is "retrograde", which means from the left to the right, spleen will be seperated at first and the pancreas will be transected later on. Secondly, only the regional lymph nodes will be dissected, which include No.10, No.11, No.18 lymph nodes, and No.9 lymph nodes should be dissected only when the lesion is in pancreatic neck. Thirdly, the transection platform is in the left side of the lesion, but transection at pancreatic neck is not mandatory. At last, the surgical plane is anterior to the left renal fascia, prerenal fascia will be preserved.
  Arms: SRPS group

SUMMARY:
Two arms RCT is design, patients with pancreatic body or tail adenocarcinoma will be randomly assigned to the Radical Antegrade Modular Pancreaticosplenectomy (RAMPS) group or Standard Retrograde Pancreatosplenectomy (SRPS) group. The primary objective is to evaluate the effect of RAMPS on the overall survival of patients with resectable body and tail pancreatic ductal adenocarcinoma. And the secondary objective is to evaluate the disease-free survival, R0 resection rate, number of retrieved lymph nodes and perioperative outcomes like postoperative complication rate, severe complications, mortality and functional recovery time between the experimental group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old;
* Resectable pancreatic body and tail ductal adenocarcinoma with both preoperative and intraoperative evaluation(refer to NCCN guideline 2018 of Pancreatic Cancer);
* ECOG Performance Status 0-1;
* Adenocarcinoma of pancreatic body and tail duct, without distant metastasis and ascites;
* The estimated survival time is ≥ 3 months;
* Follow-up in time and obey the research requirements;
* Be voluntary to this clinical trial and can sign the informed consent;
* Normal hematological index (Leukocyte, platelet, liver function, renal function, DIC, electrolyte index, Hb >10g/dL).

Exclusion Criteria:

* The patients with distant metastasis according to preoperative tumor staging;
* Patients with recurrent pancreatic ductal adenocarcinoma;
* The artery or vein is involved and could not be resected or reconstructed(according to preoperative evaluation or intraoperative evaluation after exploration);
* Patients with cardiopulmonary disfunction and cannot tolerate operation;
* The patients accepted neoadjuvant chemotherapy and radiotherapy before operation;
* Patients with other malignancies or hematopathy
* Before the operation, the total bilirubin was more than 250 μmol/L without preoperative biliary drainage or after biliary drainage, the total bilirubin was still more than 250 μmol/L;
* Pregnancy diagnosed, planned pregnancy and lactating female patients
* Refusal to sign consent.
* Intraoperative exclusion include:Tumor metastasis; not pancreatic primary disease; unresectable pancreatic body/tail adenocarcinoma
* Postoperative exclusion include: not pancreatic ductal adenocarcinoma according to pathological examination.
* Withdrawal of informed consent;
* Willingness to withdraw from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 21 months
  Overall survival was defined as the time from surgery to either death or last follow-up. Patients will be observed or contacted every 2 months in the first 2 years after surgery and then every 3 months thereafter. Overall survival measurement will be based on patient's survival status and what is the date of death if the patient is not alive.

SECONDARY OUTCOMES:
Disease free survival | 11 months
  DFS was calculated from the date of surgery to the date of recurrence or last follow-up if recurrence did not occur. Recurrence was diagnosed by imaging examination like CT, MRI, PET-CT and PET-MRI.
R0 resection rate | 1 month
  R0 resection was defined as absence of malignant cells within 1 mm from the resection margin using the Royal College of Pathologists definition. The assessment of the margin status will be done by pathologists.
retrieved lymph nodes | 1 month
  The dissected lymph nodes will be sent to pathology department and the pathologists will separate the lymph nodes and give reports about how many lymph nodes are found and if the lymph nodes are positive or negative.

OTHER OUTCOMES:
operation time in minutes | 1 day
  Operation time means "skin to skin"time (from the surgeon start to incise the skin to the last suture of the skin)
estimated blood loss in milliliters | 1 day
  Estimated blood loss will be evaluated based on the vacuum amount, gauze weight and liquid intake
postoperative pancreatic fistula in percentage | 3 months
  According to the definition of International Study Group on Pancreatic Fistula(ISGPF)
postpancreatectomy hemorrhage in percentage | 3 months
  Postpancreatectomy hemorrhage is defined by International Study Group on Pancreatic Surgery
delayed gastric emptying in percentage | 3 months
  Delayed gastric emptying is defined by International Study Group on Pancreatic Surgery
Surgical site infection in percentage | 3 months
  Surgical site infections are defined by the Center for Disease Control and Prevention (CDC) definition, and diagnosed by positive pathogen culture in 2 weeks from surgery
30-day mortality in percentage | 1 month
  Any death within 30 days in postoperative period will be calculated
90-day mortality in percentage | 3 months
  Any death within 90 days in postoperative period will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided